CLINICAL TRIAL: NCT00734240
Title: Double Blind, Placebo-Controlled, Dose-Escalation, Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of ISIS 353512 Administered Intravenously and Subcutaneously to Healthy Volunteers
Brief Title: Safety and Tolerability of Single and Multiple Doses of ISIS 353512 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Collaborators: Anapharm (Industry)
Responsible Party: Isis Pharmaceuticals, Inc., Isis Pharmaceuticals, Inc.
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: ISIS 353512 CS1
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2010-07

CONDITIONS: Inflammatory Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (16):
- A (Experimental): single-dose cohort (n=4, randomized 3 active : 1 placebo) receiving ISIS 355312 or placebo
  Interventions: Drug: ISIS 353512
- B (Experimental): single-dose cohort (n=4, randomized 3 active : 1 placebo) receiving ISIS 353512 or placebo
  Interventions: Drug: ISIS 353512
- C (Experimental): single-dose cohort (n=4, randomized 3 active : 1 placebo) receiving ISIS 353512 or placebo
  Interventions: Drug: ISIS 353512
- AA (Experimental): multiple-dose cohort (n=4, randomized 3 active : 1 placebo) receiving 353512 or placebo
  Interventions: Drug: ISIS 353512
- BB (Experimental): multiple-dose cohort (n=4, randomized 3 active : 1 placebo) receiving ISIS 353512 or placebo
  Interventions: Drug: ISIS 353512
- CC (Experimental): multiple-dose cohort (n=4, randomized 3 active : 1 placebo) receiving ISIS 353512 or placebo
  Interventions: Drug: ISIS 353512
- G (Experimental): single-dose cohort (n=4, randomized 3 active : 1 placebo) receiving ISIS 353512 or placebo
  Interventions: Drug: ISIS 353512
- H (Experimental): single-dose cohort (n=4, randomized 3 active : 1 placebo) receiving ISIS 353512 or placebo
  Interventions: Drug: ISIS 353512
- I (Experimental): single-dose cohort (n=4, randomized 3 active : 1 placebo) receiving ISIS 353512 or placebo
  Interventions: Drug: ISIS 353512
- GG (Experimental): multiple-dose cohort (n=4, randomized 3 active : 1 placebo) receiving ISIS 353512 or placebo
  Interventions: Drug: ISIS 353512
- HH (Experimental): multiple-dose cohort (n=4, randomized 3 active : 1 placebo) receiving ISIS 353512 or placebo
  Interventions: Drug: ISIS 353512
- II (Experimental): multiple-dose cohort (n=4, randomized 3 active : 1 placebo) receiving ISIS 353512 or placebo
  Interventions: Drug: ISIS 353512
- F (100 mg) (Experimental): single-dose cohort (n=4, randomized 3 active: 1 placebo) receiving ISIS 353512 or placebo
  Interventions: Drug: ISIS 353512
- Dose-Titration 1 (Experimental): multiple-dose cohort (n=4, randomized 3 active: 1 placebo) receiving ISIS 353512 or placebo
  Interventions: Drug: ISIS 353512
- F (200 mg) (Experimental): single-dose cohort (n=4, randomized 3 active: 1 placebo) receiving ISIS 353512 or placebo
  Interventions: Drug: ISIS 353512
- Dose-Titration 7 (Experimental): multiple-dose cohort (n=4, randomized 3 active: 1 placebo) receiving ISIS 353512 or placebo
  Interventions: Drug: ISIS 353512

INTERVENTIONS:
Drug: ISIS 353512 — 50 mg via 2 hour IV infusion, single dose
  Arms: A
Drug: ISIS 353512 — 50 mg via 2 hour IV infusion, 6 doses over 22 days
  Arms: AA
Drug: ISIS 353512 — 50 mg via SC injection, single dose
  Arms: G
Drug: ISIS 353512 — 50 mg via SC injection, 6 doses over 22 days
  Arms: GG
Drug: ISIS 353512 — 2 hour IV infusion, 50 mg on day 3, 100 mg on day 5, and 200 mg on day 8
  Arms: Dose-Titration 1
Drug: ISIS 353512 — 100 mg via 2 hour IV infusion, single dose
  Arms: B
Drug: ISIS 353512 — 200 mg via 2 hour IV infusion, single dose
  Arms: C
Drug: ISIS 353512 — 100 mg via SC injection, single dose
  Arms: H
Drug: ISIS 353512 — 200 mg via SC injection, single-dose
  Arms: I
Drug: ISIS 353512 — 100 mg via 2 hour IV infusion, 6 doses over 22 days
  Arms: BB
Drug: ISIS 353512 — 200 mg via 2 hour IV infusion, 6 doses over 22 days
  Arms: CC
Drug: ISIS 353512 — 100 mg via SC injection, 6 doses over 22 days
  Arms: HH
Drug: ISIS 353512 — 200 mg via SC injection, 6 doses over 22 days
  Arms: II
Drug: ISIS 353512 — 100 mg via SC injection PLUS an oral treatment of a NSAID, acetaminophen, or oral placebo
  Arms: F (100 mg)
Drug: ISIS 353512 — 200 mg via SC injection PLUS an oral treatment of a NSAID, acetaminophen, or steroid
  Arms: F (200 mg)
Drug: ISIS 353512 — 2 hour IV infusion, 50 mg on day 1, 100 mg on day 3, 100 mg on day 5 and 200mg on day 8
  Arms: Dose-Titration 7

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single and multiple doses of ISIS 353512, to evaluate the blood concentration and rate elimination of ISIS 353512 from the blood, and to evaluate the effectiveness of ISIS 353512 in lowering a protein in the blood associated with inflammation.

DETAILED DESCRIPTION:
This will be a Phase 1, double blind, placebo-controlled, dose-escalation study conducted at a single center to 1)evaluate the safety and tolerability of single and multiple doses of ISIS 353512 administered intravenously and subcutaneously, 2)evaluate the pharmacokinetic profile of single and multiple doses of ISIS 353512 administered intravenously and subcutaneously, and 3)evaluate the pharmacodynamics of ISIS 353512 in lowering constitutive levels of c-reactive proteins in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55 years
* Male or female although females must be post-menopausal or surgically sterile
* In good health
* BMI < 32 kg/m2
* Give written informed consent to participate in the study
* hsCRP at Screening ≥ 0.50 mg/L and ≤ 5.0 mg/L (for 2 measurements ≥ 2 weeks apart; with difference between measurements ≤ 2.5 mg/L)(Multiple Dose Subjects only, not including dose-titration cohorts)

Exclusion Criteria:

* Pregnant women, nursing mothers or women of childbearing potential
* Clinically significant abnormalities in medical history or physical examination
* Clinically significant ECG abnormalities or vital sign abnormalities (systolic blood pressure < 90 mm Hg or > 140 mm Hg, diastolic blood pressure < 50 mm Hg or > 90 mm Hg or heat rate < 50 or > 100 bpm) at Screening
* Clinically significant abnormalities on laboratory examination, other than hsCRP
* Clinically significant abnormalities in coagulation parameters
* Positive test for HIV, TB (PPD test) or hepatitis B or C at Screening
* History of latent or active tuberculosis or exposure to endemic areas within 8 weeks prior to PPD test at Screening
* History of positive PPD test or positive PPD test result (≥ 5 mm) indicating possible tuberculosis infection
* Fasting triglycerides > 400 mg/dL at Screening
* Malignancy (with the exception of basal or squamous cell carcinoma of the skin if adequately treated and no recurrence for > 1 year)
* Evidence of ongoing chronic inflammatory condition or infection
* Any other concurrent condition which, in the opinion of the Investigator, would preclude participation in this study or interfere with compliance
* Regular use of alcohol within 6 months prior to Screening (> 14 units of alcohol per week; 1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol)
* Use of soft drugs (such as marijuana) within 3 months prior to Screening or hard drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to Screening, or positive urine drug screen at Screening
* Smoking > 10 cigarettes per day
* Use of an investigational drug or participation in an investigational study involving a small molecule with 30 days prior to dosing or participation in an investigational study involving biologic compounds within 90 days prior to dosing
* Regularly taking OTC medications and/or vitamin supplements that may alter CRP, e.g., NSAIDs, aspirin, vitamin E, fish oil, within 14 days prior to Screening
* Receiving prescription medications, including hormone replacement therapy, statins, TNF-α inhibitors, or other anti-inflammatory or immunosuppressive drugs within 30 days prior to Screening
* Immunization with a live attenuated vaccine one month prior to dosing or planned vaccination during the course of the study
* Blood donation of 50 to 499 mL within 30 days of Screening or of > 499 mL within 60 days of Screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2008-07; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single and multiple doses of ISIS 353512 administered intravenously and subcutaneously. | 14 Days post treatment of each cohort

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic profile of single and multiple doses of ISIS 353512 administered intravenously and subcutaneously. | 14 Days post treatment of each cohort
To evaluate the pharmacodynamics of ISIS 353512 administered intravenously and subcutaneously. | 14 Days post treatment of each cohort

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, M.D., Principal Investigator — Anapharm
Locations (1):
- Anapharm, Montreal, Quebec, Canada